CLINICAL TRIAL: NCT04987645
Title: Randomized Controlled Trial Comparing the Impact of Water Assisted Colonoscopy vs Air Insufflation on Resident Training
Brief Title: Impact of Water Assisted Colonoscopy vs Air Insufflation on Resident Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Maria MacDonald, Medical Student, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021.161
Record Dates: First submitted 2021-07-20; First posted 2021-08-03 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Water Assisted Colonoscopy

STUDY DESIGN:
Intervention Model Description: Each participant would be randomly assigned to either water only or water and air insufflation on insertion via a computer-generated random number.
Who Masked: Participant
Masking Description: The participant will be blinded to the intervention until after the pain score has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water-Assisted Colonoscopy (Other): If this intervention is chosen randomly, the trainee will use water only technique for insertion.
  Interventions: Procedure: Water-only infusion technique
- Water and Air Insufflation (Other): If this intervention is chosen randomly, the trainee will use water and air insufflation technique for insertion.
  Interventions: Procedure: Water infusion and air insufflation

INTERVENTIONS:
Procedure: Water-only infusion technique — During a routine colonoscopy, a resident in the study will use water only infusion technique for this intervention. This intervention is used to look at the impact that water assisted colonoscopy has on resident learning.
  Arms: Water-Assisted Colonoscopy
Procedure: Water infusion and air insufflation — During a routine colonoscopy, a resident in the study will use water infusion and air insufflation technique for this intervention. This intervention is used to look at the impact that water assisted colonoscopy has on resident learning.
  Arms: Water and Air Insufflation

SUMMARY:
This study will be a randomized trial comparing the use of only water or water and air insufflation during colonoscopy insertion by trainees. This study will be looking at the impact that water-assisted colonoscopy has on resident learning. The investigators hypothesize that the use of water only compared to water and air will improve the learning experience for trainees.

DETAILED DESCRIPTION:
In this trial, the investigators will offer participation in the study when patients present for their scheduled routine colonoscopy. The participants will be asked to give consent for the colonoscopy procedure and participation in the trial. After consent is obtained and information is taken from the participants, each participant would be randomly assigned to either water only or water and air insufflation on insertion via a computer-generated random number. All patients over the age of 18 presenting for their scheduled colonoscopy at either the Health Sciences Centre or St. Clare's Mercy Hospital in St. John's, Newfoundland, can participate in the study. The colonoscopy will then be done in the usual manner with appropriate sedation. Patients will then be debriefed regarding their colonoscopy following the procedure in recovery. At the completion of the data extraction above, all trainee participants will undergo a semi-structured exit interview with one of the study investigators.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 presenting for their scheduled routine colonoscopy at either the Health Sciences Center or St. Clare's Mercy Hospital in St. John's, NL, can participate in the study.

Exclusion Criteria:

* Previous bowel resection, refusal to participate, inability to provide informed consent, known bowel obstruction, emergency colonoscopy. It will be noted if patients have had a previous hysterectomy, patient's age, BMI, gender, and quality of bowel preparation as these factors have been known to prolong cecal intubation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Cecal Intubation Rate | Cecal intubation rate with a 12-15 minute time limit before staff takes over
  The percentage of success in which the trainee advances the colonoscope to the cecum.

SECONDARY OUTCOMES:
Time to transverse colon intubation | Time from the start of the colonoscopy until the trainee reaches the transverse colon.
  The time it takes for the trainee to insert the colonoscope to intubate the transverse colon.
Patient comfort | Recorded during the colonoscopy
  Nurse Assessed Patient Comfort Score will be used to assess patient comfort.
Sedation dosage required | Duration of the colonoscopy
  We will document how much sedation was required during the procedure. A standard dosage will be given to all patients at the start of the procedure. If more sedation was needed during the procedure, this will be recorded.
Semi-structured exit interview | After the data extraction (five minutes to complete)
  At the completion of the data extraction, all trainee participants will undergo a semi-structured exit interview with one of the study investigators to assess their learning experience.
Rate of transverse colon intubation | Time from colonoscope insertion to transverse colon intubation.
  The percentage of success in which the trainee advances the colonoscope to the transverse colon.
Polyp/adenoma detection rate | This will occur after all the procedures have been completed. Will take roughly 1-2 days to record the number of polpys/adenomas detected.
  After the procedures are completed, a study investigator will review the Meditech records and record the number of polyps/adenomas detected for each case.
Complications during the procedure | Any complications that take place within the time frame of the procedure will be recorded.
  Any complications during the procedure will be recorded.These include bleeding, perforation resulting in subsequent abdominal surgery, and an adverse reaction to any anaesthetics used during the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Centre, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsieh YH, Koo M, Leung FW. A patient-blinded randomized, controlled trial comparing air insufflation, water immersion, and water exchange during minimally sedated colonoscopy. Am J Gastroenterol. 2014 Sep;109(9):1390-400. doi: 10.1038/ajg.2014.126. Epub 2014 Jun 3. PMID 24890443
- [Background] Lee SH, Park YK, Lee DJ, Kim KM. Colonoscopy procedural skills and training for new beginners. World J Gastroenterol. 2014 Dec 7;20(45):16984-95. doi: 10.3748/wjg.v20.i45.16984. PMID 25493011
- [Background] Leung CW, Kaltenbach T, Soetikno R, Wu KK, Leung FW, Friedland S. Water immersion versus standard colonoscopy insertion technique: randomized trial shows promise for minimal sedation. Endoscopy. 2010 Jul;42(7):557-63. doi: 10.1055/s-0029-1244231. Epub 2010 Jun 30. PMID 20593332
- [Background] Hu D, Xu Y, Sun Y, Zhu Q. Water infusion versus air insufflation for colonoscopy: a meta-analysis of randomized controlled trials. Tech Coloproctol. 2013 Oct;17(5):487-96. doi: 10.1007/s10151-013-1023-x. Epub 2013 May 8. PMID 23652813